CLINICAL TRIAL: NCT00843167
Title: Sulforaphane: A Dietary Histone Deacetylase (HDAC) Inhibitor in Ductal Carcinoma in Situ (DCIS)
Brief Title: Broccoli Sprout Extract in Treating Women Who Have Had a Mammogram and Breast Biopsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jackie Shannon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000634111; R21CA132236 (NIH); P30CA069533 (NIH); OHSU-4702 (Other: OHSU IRB)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2015-02-24 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2015-10

CONDITIONS: Breast Cancer; Precancerous Condition
Keywords: mammography; biopsy; ductal breast carcinoma in situ; atypical ductal breast hyperplasia
MeSH Terms: conditions — Breast Neoplasms; Precancerous Conditions; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulforaphane Supplement (Experimental): Patients receive oral broccoli sprout extract supplementation three times daily for 2-8 weeks in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: broccoli sprout extract
- Placebo (Placebo Comparator): Patients receive oral placebo supplementation three times daily for 2-8 weeks in the absence of unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: broccoli sprout extract — Given orally
  Arms: Sulforaphane Supplement
Other: placebo — Given orally
  Arms: Placebo

SUMMARY:
RATIONALE: Broccoli sprout extract supplements may slow the growth of tumor cells or abnormal cells and may be an effective treatment for ductal carcinoma in situ and/or atypical ductal hyperplasia.

PURPOSE: This randomized phase II trial is studying how well broccoli sprout extract works in treating women with a diagnosis of breast cancer, ductal carcinoma in situ and/or atypical ductal hyperplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the correlation between supplemental sulforaphane (broccoli sprout extract) dose and concentrations of sulforaphane and its metabolites in blood and urine samples from women positive for cancer, ductal carcinoma in situ and/or atypical ductal hyperplasia.
* To determine the effect of this supplement on biomarkers of prognosis in these patients.
* To determine the effect of this supplement on HDAC inhibition in peripheral blood cell and normal and cancerous breast tissue samples from these patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Sulforaphane Supplement: Patients receive oral broccoli sprout extract supplementation three times daily for 2-8 weeks in the absence of unacceptable toxicity.
* Placebo: Patients receive oral placebo supplementation three times daily for 2-8 weeks in the absence of unacceptable toxicity.

Blood and urine samples are collected at baseline and after completion of study treatment for laboratory biomarker studies. Patients scheduled to undergo surgery (mastectomy or lumpectomy) also undergo breast tissue sample collection at baseline and at the time of surgery. Samples are analyzed for sulforaphane metabolism (isothiocyanate levels), HDAC activity (acetylated histone expression), cell proliferation (Ki-67 index by IHC), and apoptosis (TUNEL assay).

Patients complete questionnaires at baseline and periodically during study about their dietary history, family history, cruciferous vegetable intake, adverse events, and dietary and medication changes.

After completion of study therapy, patients are followed at/around 30 days.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnostic mammogram
* English speaking

EXCLUSION CRITERIA:

* Pregnancy (as determined by urine human chorionic gonadotropin (hCG) test)
* No biopsy referral after diagnostic mammogram
* Patient reported breast feeding
* Significant active medical illness which in the opinion of the investigator would preclude protocol treatment
* History of or active liver disease or baseline total bilirubin greater than institutional upper limit of normal
* Patient reported allergy or sensitivity to cruciferous vegetables
* Use of oral antibiotics within three months prior to randomization
* Oral steroid therapy at enrollment
* Current therapy with valproate acid or SAHA
* Current use of nutrient supplements or herbal remedies containing sulforaphane and unwillingness or inability to quit 72 hours prior to randomization and for the duration of the trial
* Radiation for currently-diagnosed disease prior to or during study supplementation
* Chemotherapy for currently-diagnosed disease prior to or during study supplementation

Ages: 21 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Atwell LL, Zhang Z, Mori M, Farris P, Vetto JT, Naik AM, Oh KY, Thuillier P, Ho E, Shannon J. Sulforaphane Bioavailability and Chemopreventive Activity in Women Scheduled for Breast Biopsy. Cancer Prev Res (Phila). 2015 Dec;8(12):1184-1191. doi: 10.1158/1940-6207.CAPR-15-0119. Epub 2015 Oct 28. PMID 26511489
- [Derived] Zhang Z, Atwell LL, Farris PE, Ho E, Shannon J. Associations between cruciferous vegetable intake and selected biomarkers among women scheduled for breast biopsies. Public Health Nutr. 2016 May;19(7):1288-95. doi: 10.1017/S136898001500244X. Epub 2015 Sep 2. PMID 26329135

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This clinical trial was conducted between 12/23/2008 to 3/27/2013 at Oregon Health and Science University's (OHSU) Center for Women's Health Breast Center in Portland, OR. English-speaking women were recruited to participate in the study based on the following inclusion criteria: ≥ 21 years, diagnostic mammogram with results that require biopsy.
Period: Treatment Period
Arm/Group | Sulforaphane Supplement | Placebo
Started | 27 | 27
Completed | 24 | 19
Not Completed | 3 | 8
Not completed — Adverse Event | 1 | 5
Not completed — Withdrawal by Subject | 2 | 3
Period: Follow-up
Arm/Group | Sulforaphane Supplement | Placebo
Started | 24 | 24
Completed Final Visit | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulforaphane Supplement | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 18 | 42
  >=65 years | 3 | 9 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.5) | 55.3 (14.3) | 54.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 26 | 24 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Isothiocyanate in Urine Samples as Assessed at Baseline and After Completion of Study Therapy
Description: Isothiocyante including sulforaphane in micromolar (µM) concentration was measured following standard chemical measurement procedures and divided by the creatinine values in millimolar (mM) concentration.
Time Frame: Baseline and end of study (up to 8 weeks)
Measure: Mean (Standard Error); unit: µM/mM creatinine
Arm/Group | Sulforaphane Supplement | Placebo
Number analyzed (Participants) | 27 | 27
µM/mM creatinine | 1.00 (0.334) | -0.05 (0.02)

2. Primary Outcome: Change in Ki-67 as Assessed at Baseline and After Completion of Study Therapy
Description: Ki-67 was measured through immunohistochemistry method. A modified H-score was recorded, which involved semi-quantitative assessment of both staining intensity (graded as 1-3 with 1 representing weak staining, 2 moderate staining, and 3 strong staining) and percentage of positive cells. The range of the H-score was 0-300. The maximum score indicates the strongest expression, the minimum score indicates no expression of positive tumor area.
Time Frame: Baseline and end of study (up to 8 weeks)
Population: Maximum two observations (pre- and post- treatments) were expected per participant. Linear mixed effect models were used to calculate adjusted least square means (LSMEANS) and 95% confidence intervals,& to test the statistical significance of the difference between pre- and post- treatments within each group, as well as between treatment groups.
Measure: Least Squares Mean (95% Confidence Interval); unit: Log 2 (H-score)
Groups:
- Benign Tissue; Ki-67: Sulforaphane Supplement = 23, Placebo = 25
- DCIS Tissue; Ki-67: Sulforaphane Supplement= 6, Placebo = 13
- Invasive Ductal Carcinoma Tissue; Ki-67: Sulforaphane Supplement= 7, Placebo= 6
Arm/Group | Benign Tissue; Ki-67 | DCIS Tissue; Ki-67 | Invasive Ductal Carcinoma Tissue; Ki-67
Number analyzed (Participants) | 48 | 19 | 13
Log 2 (H-score)
  Sulforaphane Supplement | -1.39 [-2.23 to -0.55] | 0.42 [-1.18 to 2.02] | 0.98 [-3.89 to 5.85]
  Placebo | 0.23 [-0.61 to 1.07] | -0.48 [-1.69 to 0.72] | 0.28 [-3.22 to 3.78]

3. Primary Outcome: Change in Histone Deacetylase (HDAC) Activity as Assessed in Peripheral Blood Mononuclear Cells (PBMC) at Baseline and After Completion of Study Therapy
Description: PBMC HDAC activity was evaluated using the positive control, sodium butyrate.HDAC activity is expressed relative to PBMC protein content and negative control.
Time Frame: Baseline and End of Study (up to 8 weeks)
Population: PBMCs available pre-/post-intervention.
Measure: Mean (Standard Error); unit: pmol/min/mg protein
Arm/Group | Sulforaphane Supplement | Placebo
Number analyzed (Participants) | 23 | 24
pmol/min/mg protein | -80.39 (48.53) | 27.52 (32.58)

4. Secondary Outcome: Treatment Compliance
Description: For treatment compliance, participants who take >=80% of the prescribed pills will be considered to be treatment-compliant.
Time Frame: Baseline and end of study (up to 8 weeks)
Measure: Number; unit: participants
Groups:
- Treatment: Patients receive oral placebo supplementation three times daily for 2-8 weeks in the absence of unacceptable toxicity.
  placebo: Given orally
Arm/Group | Sulforaphane Supplement | Treatment
Number analyzed (Participants) | 27 | 27
participants | 19 | 16

ADVERSE EVENTS:
Arm/Group | Sulforaphane Supplement | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 8/27 | 9/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulforaphane Supplement (N=27) | Placebo (N=27)
Bloating (Gastrointestinal disorders) | 5 | 5
Gas/Flatulence (Gastrointestinal disorders) | 1 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 2
Nausea/Vomiting (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Taste Alteration (Nervous system disorders) | 0 | 2
Bruising (Musculoskeletal and connective tissue disorders) | 1 | 1
Tingling tongue sensation (Nervous system disorders) | 0 | 1
Feeling tired (Psychiatric disorders) | 0 | 1 — The participant thinks it might be due to stress or these pills
More sleep (Nervous system disorders) | 0 | 1
Sleeping less (Nervous system disorders) | 0 | 1
Insomnia (Nervous system disorders) | 0 | 1
Arthritic pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Allergy (Immune system disorders) | 0 | 1
Cramping (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Heartburn (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No